CLINICAL TRIAL: NCT05955534
Title: A Multicenter, Randomized Controlled Trial of Concomitant Bedside Percutaneous Tracheostomy and Ultrasound Gastrostomy
Brief Title: Concomitant Bedside Percutaneous Tracheostomy and Ultrasound Gastrostomy
Acronym: TPUG
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of supporting resources
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Richard Gentry Wilkerson, Associate Professor, Director of Clinical Research, Assistant Residency Program Director, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00104764
Record Dates: First submitted 2023-06-28; First posted 2023-07-21 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Gastrostomy; Ventilatory Failure; Respiratory Failure
Keywords: Ventilator Dependent Respiratory Failure; Tracheostomy and Percutaneous Ultrasound Gastrostomy (TPUG); Percutaneous Radiologic Gastrostomy (PRG); PEG; Percutaneous Endoscopic Gastrostomy; Tracheostomy; Gastrostomy
MeSH Terms: conditions — Hypoventilation; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: All patients enrolled will receive bedside tracheostomy, but each patient will be randomly assigned a common method for gastrostomy placement. Patients in the control group will receive a bedside tracheostomy along with a common method of gastrostomy placement other than PUG, which may be performed at the same time or at a different time in relation to the tracheostomy. Patients in the intervention group will receive a bedside tracheostomy and a PUG at the same time using an FDA-cleared device.
Who Masked: Investigator
Masking Description: Participants will be randomly assigned to either the intervention group (TPUG) or the control group using a 1:1 randomization scheme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Group (Placebo Comparator): The control group will receive percutaneous bedside tracheostomy along with gastrostomy methods other than PUG, including but not limited to Percutaneous Endoscopic or Radiologic Gastrostomy (PEG or PRG, respectively), or surgical gastrostomy.
  Interventions: Procedure: PEG; Procedure: PRG
- Intervention Group (TPUG) (Experimental): The intervention group will receive concomitant percutaneous bedside tracheostomy and PUG.
  Interventions: Device: TPUG

INTERVENTIONS:
Device: TPUG — Tracheostomy shall utilize any FDA approved device for the performance of percutaneous dilatational tracheostomy. PUG shall be performed using the only FDA-cleared device for ultrasound gastrostomy, the PUMA-G System.
  Other Names: Percutaneous Tracheostomy and Percutaneous Ultrasound Gastrostomy
  Arms: Intervention Group (TPUG)
Procedure: PEG — Each site will perform the procedures of gastrostomy placement using the devices according to their institutional policy and guidelines.
  Other Names: Percutaneous Endoscopic Gastrostomy
  Arms: Control Group
Procedure: PRG — Each site will perform the procedures of gastrostomy placement using the devices according to their institutional policy and guidelines.
  Other Names: Percutaneous Radiographic Gastrostomy
  Arms: Control Group

SUMMARY:
The goal of this research study is to assess the FDA approved technique for inserting a feeding tube (gastrostomy) along with a breathing tube (tracheostomy) for patients that cannot breathe or eat on their own in the ICU (Intensive Care Unit). All subjects in the study will receive a tracheostomy, but each patient will be randomly assigned a common method for gastrostomy placement. The placement of the tube and tracheostomy will occur as part of normal clinical practice. Researchers will compare subjects in the control group and the intervention group to evaluate the benefits of performing a tracheostomy and gastrostomy tube at the same time. Researchers will also evaluate the likelihood of the PUG procedure decreasing a patient's length of stay in the ICU.

DETAILED DESCRIPTION:
The research team will assess eligibility during the screening period for percutaneous tracheostomy and gastrostomy. Once eligibility is assessed, participants and/or their legally authorized representative (LAR) will be approached for consent and enrollment into the trial. Randomization occurs at the time of the subject's enrollment, and participants will be randomized to either the Control or Intervention (TPUG) groups using randomly assigned numbers. The study team will also be blinded to the assigned group prior to recruitment to limit selection bias. The intervention group will receive concomitant placement of the tracheostomy and PUG, which will be performed using the FDA-cleared device for ultrasound gastrostomy, the PUMA-G System. The control group will receive percutaneous bedside tracheostomy along with gastrostomy methods other than PUG. Each site will perform the procedures of tracheostomy and gastrostomy using the devices according to their institutional policy and guidelines. Investigators will utilize case report forms (CRFs) and chart review to collect demographic information, important medical events, illnesses, and laboratory data needed for outcomes assessment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent must be obtained from the participant or a Legally Authorized Representative before any trial-specific assessment is performed
* Male or female ≥ 18 years of age
* Participants with Ventilator Dependent Respiratory Failure (VDRF)
* Indication for a bedside percutaneous tracheostomy procedure using an FDA approved percutaneous dilatational tracheostomy device
* Indication for percutaneous gastrostomy including Percutaneous Ultrasound (PUG), Percutaneous Radiologic (PRG), and Percutaneous Endoscopic Gastrostomy (PEG) using an FDA approved gastrostomy kit
* No contraindications to bedside percutaneous tracheostomy OR gastrostomy
* Women of childbearing potential must have negative serum or urine pregnancy test during the current hospitalization

Exclusion Criteria:

* History of prior gastrostomy, tracheostomy, laryngectomy, gastrostomy prior to tracheostomy decision, known head and neck and gastrointestinal abnormality (cancer, congenital abnormality, anatomic variants).
* Hospitalization > 21 days at the time of screening
* Known social discharge issues that in the opinion of the investigator will substantially impact the LOS.
* Participants with non-survivable injuries or disease, anticipated life expectancy < 30 days.
* Uncontrolled coagulopathy
* Contraindications for percutaneous gastrostomy procedures
* Severe Ascites
* Abdominal wall infection at selected site of procedure
* Severe gastroparesis
* Gastric outlet obstruction
* Absolute contraindications to percutaneous dilatational tracheostomy procedure
* Cervical instability
* Infection at the planned insertion site
* Relative contraindications to percutaneous dilatational tracheostomy deemed present by the clinical team
* Difficult anatomy (e.g., short neck, morbid obesity, minimal next extension, or tracheal deviation)
* Severe respiratory disease resulting in inability to withstand periods of apnea or in the loss of positive pressure ventilation
* Pregnancy
* Incongruent goals of care between care team and LAR (family representative).
* Other procedure related concerns by the primary team that would affect safety of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Length of stay in ICU | ICU discharge - up to 24 weeks
  To compare the ICU (Intensive Care Unit) length of stay (days) from the time the decision is made to place a tracheostomy tube and gastrostomy tube to the time of discharge from the ICU for participants receiving TPUG versus a control group.

SECONDARY OUTCOMES:
Length of hospital stay | Hospital discharge - through study completion, an average of 45 days
  To compare the hospital length of stay (days) and total hospital costs (United States Dollars) from the time the decision is made to place a tracheostomy tube and gastrostomy tube to the time of discharge from the hospital for participants receiving TPUG versus a control group.
Demographics | End of study comparison - through study completion, an average of 45 days
  To assess confounding variables and differences between groups that could affect outcomes:
  1. Age (categorized as <50 yrs., 51-70 yrs., >70 yrs)
  2. Gender (Assigned at birth)
  3. Race (Self-Reported)
  4. Insurance (categorized as Insured versus Uninsured)
  5. Covid status (categorized as Positive, Negative, Indeterminate)
  6. Primary diagnosis
  7. Primary ICU type
  8. Charlson Score
  9. SAPS Score

CONTACTS AND LOCATIONS:
Overall Officials: Dana Beach, RN, Study Chair — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Systems, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The Principal Investigator will centrally aggregate and maintain screening and recruitment information from all study sites and routinely inform and share this data with the entire study team in a deidentified fashion. The principal investigator and co-investigators will maintain a personal participant identification list (participant numbers with the corresponding participant names) to enable records to be identified.
  The University of Maryland School of Medicine's research team will ensure that all study-related documents are collected and maintained.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Until the end of the study. Essential documents will be retained for at least 2 years.
Access Criteria: All study team members will attend online trainings to receive instruction on the protocol, consent process and associated regulatory requirements for the conduct of Clinical Trials/Human Subjects Research. All persons assisting with the trial are adequately informed about the protocol, any amendments to the protocol, any changes to the informed consent form, the trial treatments, eligibility criteria and their trial related duties and functions.